CLINICAL TRIAL: NCT05539313
Title: The Investigation and Analysis of Atria of Patients With Non-paroxysmal Atrial Fibrillation Using High-desnity Mapping and Cardiac Magnetic Resonance Imaging
Brief Title: Examination of Fibrillation Atria Using Magnetic Resonance Imaging and Endocardial High-density Mapping
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Pavel Osmancik, head of the department of arrhythmias, Charles University, Czech Republic
Other Study IDs: MRI Octarey
Record Dates: First submitted 2022-09-10; First posted 2022-09-14 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; catheter ablation; cardiac magnetic resonance; high-density mapping
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: High-density mapping — Patients will undergo magnetic resonance imaging of both atria, and interventional high-density mapping of both atria.

SUMMARY:
Cather ablation of non-paroxysmal atrial fibrillation is less effective compared to paroxysmal atrial fibrillation. Therefore, new techniques have been developed, such as high-density mapping to determine areas of focal and rotational activities. The aim is to assess the clinical efficacy of ablation focal and rotational activities, and to assess the relation between the areas of focal and rotational activities with fibrosis of both atria assessed using magnetic resonance.

DETAILED DESCRIPTION:
Pateints with non-paroxysmal atrial fibrillation will be enrolled. Before the procedure, cardiac magnetic resonance will be done to determine the extent and location of atrial fibrosis of both atria using dedicated software. The procedure itself will be done standardly, in alangosedation, from both femoral veins, using 10-pole catheter in the coronary sinus, intracardiac echocardiography, and two transseptal punctures by means of SL1 sheaths. Octarey mapping catheter (Biosense Webster, USA) wil be inserted in the left atrium, and during ongoing atrial fibrillation, a maping of left atrium will be done to locate the areas of focal and rotational activities. Afterthat, using Smart Touch ablation catheter (Biosense Webster, USA), pulmonary vein isolation will be done. When PVI is achieved, all areas of focal and rotational activities determined by high-density mapping will be performed. If sinus rhythm is achieved, the procedure is finished. If atrial fibrilaltion is organized to regular atrial, this regular tachacardia is mapped, ablated and the procedure is finished. If atrial fibrilaltion continues, mapping of the righ atrium using the same technique is done followed by catheter ablation of areas of focal and rotational activities. If atrial fibrillation is still present after all these ablation, electrical cardioversion will be done.

Patients will be discharged on following day. 5-day Holter recording will be done in 3, 6, and 12 months during standard out-patient controls.

The aim is to compare the findings of high-density mapping with findings on atrial MRI (relation between fibrosis on MRI and locations of rotational and focal activities). Furher aim is to assess the efficaccy of this kidn of ablation, i.e. the sinus rhythm maintenance in 3,6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* non-paroxysmal atrial fibrillation

Exclusion Criteria:

* creatinine > 120 umol/l
* claustrofobia
* pregnancy
* mechanical valve
* significant valve disease
* left ventricular dysfunction, EF less than 35%

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with non - paroxysmal, i.e. persistent or long-lasting persistent symptomatic atrial fibrillation fulfilling standard criteria for catheter ablation
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Sinus rhythm maintenance | 1 year
  The freedom from atrial fibrillation
MRI and high-density relation | 3 days
  The relation between areas of location and rotational activities with atrial fibrosis location

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiocenter, 3rd Medical School, Charles University and University Hospital Kralovske Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Protocol will shared after study initiation
Supporting Information: Study Protocol